CLINICAL TRIAL: NCT01266135
Title: Randomized, Double-blind, Placebo-controlled, Multiple-dose, Exploratory Proof of Concept Study to Assess the Safety, Tolerability, Efficacy, Pharmacodynamic (PD) and Pharmacokinetics of QAX576 in Patients With Rapidly Progressive IPF
Brief Title: Safety and Efficacy of QAX576 in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CQAX576A2203; 2010-020688-18
Record Dates: First submitted 2010-12-17; First posted 2010-12-24 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2015-04

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Interstitial Lung Disease; Usual Interstitial Pneumonia; Fibrosis,; Pulmonary Fibrosis,; Respiratory Disease,; Interstitial Lung Disease,; Biological Therapy,; Therapeutic Uses,
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Lung Diseases, Interstitial; Fibrosis; Pulmonary Fibrosis; Respiration Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Arm 1: QAX576 10 mg/kg (Experimental)
  Interventions: Drug: QAX576
- Arm 2: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QAX576 — QAX576 10 mg/kg intravenous infusion
  Arms: Arm 1: QAX576 10 mg/kg
Drug: Placebo — Placebo to QAX576 intravenous infusion
  Arms: Arm 2: Placebo

SUMMARY:
This study is designed to evaluate the safety, tolerability, pharmacokinetics and efficacy of QAX576 in patients with idiopathic pulmonary fibrosis.

ELIGIBILITY:
Inclusion criteria

* Diagnosis of Idiopathic Pulmonary Fibrosis (IPF), based on an appropriate clinical definition of IPF as detailed in the ATS/ERS/JRS/ALAT Statement: Idiopathic Pulmonary Fibrosis: Evidence-based Guidelines for Diagnosis and Management Diagnosis must be confirmed by a diagnostic HRCT or surgical lung biopsy.
* A 6-minute walk test (6MWT) distance ≥50 meters at Screening (use of supplemental oxygen allowed).

Exclusion criteria

* Smokers (use of tobacco products in the previous 3 months). Urine cotinine levels will be measured during screening for all subjects. Smokers will be defined as any subject who reports tobacco use or has a urine cotinine levels in the range defined as 'smokers' per the local lab.
* Lung residual volume > 120% predicted at Screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety, tolerability, and effect on lung function of multiple intravenous doses of QAX576 in patients with IPF | 1 year
Change in forced vital capacity (FVC) at 52 weeks as compared to baseline | 1 year
  Measure: FVC was measured using a spirometer according to American Thoracic Society / European Respiratory Society guidelines at screening and week 52 of the treatment period.
Safety and tolerability of QAX576. | 1 year
  Measure safety and tolerability as assessed by reported AEs and effects on routine laboratory evaluations.

SECONDARY OUTCOMES:
To evaluate the effect of multiple intravenous doses of QAX576 on measures of clinical efficacy | 1 year
To determine the pharmacokinetics of of QAX576 by measuring concentrations of QAX576 in blood | 1 year
Time to clinical worsening: | 1 year
  Measure: Time to clinical worsening defined as fall in FVC or Diffusing Capacity of the lung for Carbon Monoxide (DLco), lung transplant or lung disease (IPF)-related death
Exacerbation of IPF | 1 year
  Measure: Incidence of exacerbation of IPF during the study
Progression of fibrosis | 1 year
  Measure progression of fibrosis in the lungs as measured by Quantitative High Resolution Computerized Tomography (HRCT)
Pharmacokinetics of QAX576 | 1 year
  Measure concentrations of QAX576 and its metabolites in blood throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- United States (7):
  - Novartis Investigative Site, Gainesville, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, San Antonio, Texas
- United Kingdom (3):
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, London

REFERENCES:
- See also: Results for CQAX576A2203 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=11844